CLINICAL TRIAL: NCT06350682
Title: Resilient HIV Implementation Science With SGM Youths Using Evidence
Acronym: RISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Florida State University (Other)
Responsible Party: Principal Investigator, Man Charurat, Director, Division of Epidemiology and Prevention, University of Maryland, Baltimore
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: HP-00107323
Record Dates: First submitted 2024-02-20; First posted 2024-04-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthMPowerment (HMP) Delayed Access (No Intervention): Delayed access for 12 months to the HMP app, individuals will have access but it will be restricted
- HealthMPowerment (HMP) Open Access (Experimental): Full access to the HMP app
  Interventions: Behavioral: HealthMPowerment (HMP)

INTERVENTIONS:
Behavioral: HealthMPowerment (HMP) — Participants will be provided access to the status neutral platform (HMP)mobile app for 12 months exposure period or a delayed access period. The HMP is developed specific to RISE and will be adapted based off feedback from each local site via stakeholders/YABs. The HMP will encompass a range of features including a robust content management system and back end administrative dashboard, multi media resources and information center, social support features such as connections to peers and providers, interactive activities and self assessments, and flexible medication and health trackers. In addition the app will support HIV/STI test kit ordering and results portal and a gamified reward system. With real time analytics to monitor user engagement and response with the DHI we can adapt the delivery of tailored content to fit emergent HIV prevention and care challenges.
  Arms: HealthMPowerment (HMP) Open Access

SUMMARY:
The Resilient HIV Implementation Science with SGM Youths using Evidence (RISE) Clinical Research Center will use a Type 2 hybrid-effectiveness-implementation study to evaluate the effectiveness and implementation of HMP, a youth-tailored digital health platform. It is hypothesized that SGM youths in the HMP intervention group will demonstrate improved PrEP initiation and viral load suppression over 12 months compared to the delayed HMP group.

DETAILED DESCRIPTION:
RISE is a randomized control trial where participants are randomized (1:1) to either healthMPower (HMP) exposure for a 12 month period or delayed access to the HMP within 8 strata based on the serostatus group. HIV seropositive and HIV seronegative at risk, age group 15 to 17 or 18 to 24 years of age and country either Nigeria, Kenya, Malawi, or Zambia. Within the strata of serostatus, age, and country, participants will be randomly assigned to the next treatment allocation from a randomly permuted block sequencing using block size of four.

750 Participants will be randomly assigned to the HMP exposure while the other 750 participants will have delayed access to HMP. The HMP is a culturally adapted status neutral mobile app that works to address HIV prevention to care continuum (PHCC) for SGM youth at each of the CBSPs.

Participants who are delayed access for 12 months will be granted "Open access" for 12 months thereafter, when compared to participants who were provided access for 12 months then provided 12 months of access called "continued access" without other external support. Therefore, participants will either be provided access for 12 or 24 months depending on the randomization.

Primary outcome, clinical effectiveness endpoint for HIV seronegative at risk young will be the uptake of PrEP and for HIV seropositive viral load suppression. Secondary outcome, PHCC pathway characterized for HIV seronegative at risk youth such as PrEP education and continuation and for HIV seropositive HIV testing, linkage, and ART initiation.

ELIGIBILITY:
Inclusion Criteria:

* Male sex at birth
* Age 15-24 years
* Own an Android or iOS smartphone
* Had receptive or insertive sex with another man in the past 12 months
* Receiving care or prevention services at the CBSP-associated with the CRPS at the time of study.

Exclusion Criteria:

* Less than 15 years old
* Greater than 24 years old
* Inability or cognitively impaired to provide consent
* Does not own an Android or iOS smartphone.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1500 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation for HIV seronegative seropositive | 24 months
  For those HIV seronegative, initiation of pre-exposure prophylaxis (PrEP) (Oral PrEP dispensed by pharmacy or Long-acting injectable defined as receiving first dose)
Viral load suppression for HIV | 24 months
  HIV seropositive viral load suppression at 12 months of taking ART (defined as HIV viral load of less than 1,000 copies/mL)
RE-AIM | 24 months
  Implementation Effectiveness on reach (characteristics of participants enrolled), Adoption (HMP physician and client interaction), Implementation (barriers and facilitators), Maintenance (HMP immediate access group at 21-24 months) and cost effectiveness of the HMP (incremental costs effectiveness ration and net monetary benefit)

SECONDARY OUTCOMES:
HIV testing cascade | 12-24 months
  HIV self testing
PrEP continuum | 12-24 months
  PrEP education (restart/re-initiation)
HIV care and treatment continuum | 12-24 months
  For those HIV seropositive, antiretroviral treatment (ART) initiation and retention at 12 months
Implementation effectiveness | 24 months
  Study retention (participants who remained active at 24 months)

IPD SHARING:
Plan to Share IPD: No